CLINICAL TRIAL: NCT03506048
Title: A Phase 2 Study of Lenvatinib in Combination With Radioactive Iodine Therapy in Patients With Progressive RAI-Sensitive Differentiated Thyroid Cancer
Brief Title: Lenvatinib and Iodine Therapy in Treating Patients With Radioactive Iodine-Sensitive Differentiated Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study has been abandoned for lack of accrual
Sponsor: Emory University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Taofeek K. Owonikoko, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00101617; NCI-2018-00144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4271-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Differentiated Thyroid Gland Carcinoma; Thyroid Gland Follicular Carcinoma; Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (lenvatinib) (Experimental): Patients receive lenvatinib PO QD for 8 weeks and up to 12 weeks in the absence of disease progression or unaccepted toxicity. Patients also receive radioactive iodine (RAI) I-131 orally as standard of care.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Given orally once daily continuously
  Other Names: E7080; ER-203492-00; Multi-Kinase Inhibitor E7080

SUMMARY:
This phase II trial studies how well lenvatinib works when given together with standard of care iodine I-131 in treating patients with radioactive iodine-sensitive differentiated thyroid cancer. Lenvatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of lenvatinib pretreatment along with radioactive iodine (RAI) in patients with previously treated RAI sensitive thyroid cancer.

SECONDARY OBJECTIVES:

I. To demonstrate the safety of the combination of lenvatinib and RAI in patients with Iodine sensitive differentiated thyroid carcinoma (DTC).

II. To assess dynamic changes in established serum based biomarkers of DTC (thyroglobulin [Tg] and Tg antibody).

III. To explore the utility of protein and genetic biomarkers to predict treatment efficacy.

OUTLINE:

Patients receive lenvatinib orally (PO) once daily (QD) for 8 weeks and up to 12 weeks in the absence of disease progression or unaccepted toxicity. Patients also receive iodine I-131 PO daily as standard of care.

After completion of study treatment, patients are followed up within 6 weeks, every 3 months for 1 year, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Prior treatment with therapeutic dose of radioactive iodine (> 50 mCi) with evidence of RAI uptake on delayed scan and with progression (biochemical or anatomic) within 12 months of RAI
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky ≥ 80%)
* Leukocytes ≥ 3,000/µL
* Absolute neutrophil count ≥ 1,500/µL
* Platelets ≥ 100,000/µL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance ≥ 60 mL/min/1.73 m² for patients with creatinine levels above institutional normal
* Confirmed diagnosis of differentiated thyroid cancer (follicular or papillary thyroid cancer and their variants)
* Ability and willingness to use appropriate contraception; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 2 weeks after completion of lenvatinib administration
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) by chest x-ray or as ≥ 10 mm (≥ 1 cm) with computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have received RAI within 12 weeks of planned retreatment
* Prior receipt of cumulative RAI doses in excess of 1000 mCi
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1)
* Patients who are receiving any other investigational agents
* Patients with previously untreated and or symptomatic brain metastases are excluded from this clinical trial because of the risk of intracranial bleeding with angiogenic agents and tumoral swelling from RAI
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to lenvatinib
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with uncontrolled hypertension (requirement for more than 2 blood pressure [BP] medications or grade 2 or higher BP elevation while on adequate doses of not more than 2 antihypertensive agents) are excluded from the study because one of the significant adverse events of lenvatinib is worsening hypertension
* Fridericia's corrected QT (QTcF) interval prolongation greater than 500 ms
* Recent arterial thromboembolic event within the previous 6 months
* Urine dipstick proteinuria ≥ 2+ or nephrotic range proteinuria on ≥ 2 gram in 24-hour urine
* History of gastrointestinal perforation, abscess or fistula
* History of and or medical condition (e.g. diverticular disease; aneurysm) that predisposes to risk of major hemorrhage
* Pregnant women are excluded from this study because lenvatinib is a tyrosine kinase inhibitor agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenvatinib, breastfeeding should be discontinued if the mother is treated with lenvatinib
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with lenvatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek K. Owonikoko, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Lenvatinib): Patients receive 24mg of lenvatinib by mouth (PO) everyday (QD) for 8 weeks and up to 12 weeks in the absence of disease progression or unaccepted toxicity. Patients also receive radioactive iodine (RAI) I-131 orally as standard of care.
  Lenvatinib: Given orally once daily continuously
Period: Overall Study
Arm/Group | Treatment (Lenvatinib)
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Time To Progression
Description: The time-to-progression (TTP) will be the primary endpoint for study, and will be determined using all enrolled patients in accordance with the intention to treat (ITT) principle. The study is formulated to have power = 0.90 at the significance level of 0.05 to correctly detect that improvement in median time to progression from 6 moths to 12 months.
Time Frame: Up to 2 years from when a participant started at baseline
Population: No data displayed because Outcome Measure has zero total participants analyzed.The study was closed for lack of feasibility due to lack of enrollment. Therefore there is no data to report.
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 0

2. Secondary Outcome: Best Objective Response
Description: Objective response rate and disease control rate will be summarized. For the expansion cohorts, objective response rate will be presented along with 95% exact confidence intervals.
  Patients will be assigned one of the following categories: complete response (CR), partial response (PR), stable disease (SD), progressive disease, non-evaluable, and disease control (CR + PR + SD). The same method of assessment and the same technique will be used to characterize each identified and reported lesion at baseline and during follow-up.
Time Frame: Up to 2 years from when a participant started at baseline
Population: as for outcome 1
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Thyroglobulin Levels
Description: Biochemical response will be assessed using suppressed and stimulated thyroglobulin. Thyroglobulin will be checked at baseline and post RAI every 3 months for 12 months and every 4-6 months thereafter as clinically indicated. Stimulated thyroglobulin obtained at baseline, prior to RAI, at 3 months, 6 months and 12 months post RAI will be used to define biochemical response. Unstimualte Tg levels may be used if unable to obtain stimulated Tg
Time Frame: Up to 2 years from when a participant started at baseline
Population: No data displayed because Outcome Measure has zero total participants analyzed.The study was closed for lack of feasibility due to lack of enrolment. Therefore there is no data to report.
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Thyroglobulin Antibody Levels
Description: Biochemical response will be assessed using suppressed and stimulated thyroglobulin antibody. Thyroglobulin antibody will be checked at baseline and post RAI every 3 months for 12 months and every 4-6 months thereafter as clinically indicated. Stimulated thyroglobulin obtained at baseline, prior to RAI, at 3 months, 6 months and 12 months post RAI will be used to define biochemical response. Unstimualte Tg levels may be used if unable to obtain stimulated Tg
Time Frame: Up to 2 years from when a participant started at baseline
Population: as for outcome 1
Arm/Group | Treatment (Lenvatinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Arm/Group | Treatment (Lenvatinib)
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Early termination of the study because of recruitment difficulties lead to insufficient data collection and analysis of primary and secondary outcome measures. Pharmaceutical company terminated study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03506048/Prot_SAP_000.pdf